CLINICAL TRIAL: NCT02957643
Title: Treatment of Iron Defieciency Anemia
Brief Title: Substitution of the Normal Levels of Iron and Hemoglobin in Pregnant Women With Iron Supplement
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, ANGELOS DANIILIDIS, Assistant professor of obstetrics and gynaecology A.U.TH., Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HippokratioGH
Record Dates: First submitted 2016-10-12; First posted 2016-11-08 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Prevention of Anemia
MeSH Terms: interventions — Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pregnant women (Placebo Comparator): iron dosage 1 per day for 3 months
  Interventions: Drug: Iron
- pregnant women with anemia (Experimental): iron dosage 1 per day for 6 months
  Interventions: Drug: Iron

INTERVENTIONS:
Drug: Iron — oral treatment
  Other Names: oral iron

SUMMARY:
The purpose of the study is to investigate the effectiveness of iron in the treatment of iron deficiency in pregnant 2nd and 3rd quarter. Every 30 days the investigators measure the hemoglobin, hematocrit and iron in serum and assess the course of treatment.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effectiveness of iron in the treatment of iron deficiency in pregnant 2nd and 3rd quarter. Every 30 days the investigators measure the hemoglobin, hematocrit and iron in serum and assess the course of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Age more or equal of 18 years
2. Registration consent
3. Have complete 12h week of pregnancy
4. Hemoglobin levels <10,5 ptl
5. Hematocrit < 32 %

Exclusion Criteria:

1. Age <18 years
2. Absent registration consent
3. Step of pregnancy less than 12 weeks
4. Coadministration formulations iron oral or parenterally
5. Background of liver kirrosis
6. Background of aimosidirosis
7. Background acquired or chronic aimatochromatosis
8. Aplastic , Hemolytic anemia and chronic diseases
9. Chronic pancreatitis
10. Subjective renal or/and liver disease
11. Hypothyroidism or yperthyreoeidismos

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Measured and reported effectiveness of iron in the treatment of iron deficiency in pregnant 2nd and 3rd quarter with questionnaire | up to 24 months
  Measured and reported effectiveness of iron in the treatment of iron deficiency in pregnant

SECONDARY OUTCOMES:
adverse reactions | up to 24 months
  adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: PANAGIOTIS MATSOUKATIDIS, MD,Msc, Principal Investigator — Aristotle University Of Thessaloniki; CHARALABOS KOLVATZIS, MD, Principal Investigator — Aristotle University Of Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
email contact
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: up to two years upon completion
Access Criteria: email contact